CLINICAL TRIAL: NCT01436877
Title: One-arm Feasibility and Prospective Pivotal Study to Assess the Safety and Efficacy of MediTate Temporary Implantable Nitinol Device (TIND) in Subjects Presenting Bladder Outlet Obstruction Secondary to BPH
Brief Title: Assessing Safety & Efficacy of MediTate Temporary Implant in Subjects With Benign Prostate Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-01
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Bladder Neck Obstruction; Benign Prostate Hyperplasia
Keywords: BPH; bladder neck obstruction; Bladder neck obstruction secondary to BPH
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- device (Experimental): Insertion of Temporary Implantable Nitinol Device (TIND)
  Interventions: Device: Insertion of Temporary Implantable Nitinol Device (TIND)

INTERVENTIONS:
Device: Insertion of Temporary Implantable Nitinol Device (TIND) — Subjects will be inserted with the Temporary Implantable Nitinol Device (TIND) to the bladder neck and urethral prostate for 5 days and thereafter the TIND will be withdrawn in the doctor office.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MediTate Temporary Implantable Nitinol Device (TIND) used to alleviate symptoms of Bladder Outlet Obstruction (BOO) secondary to Benign Prostate Hyperplasia (BPH).The TIND is inserted in the bladder neck and prostatic urethra under local anesthesia for few days and taken out some 5 days later in the doctors office.

ELIGIBILITY:
Inclusion Criteria:

Main IC:

* Subject signed informed consent prior to the performance of any study procedures.
* Male with BPH, who are at least 50 years of age and that were diagnosed with BOO.
* IPSS symptom severity score ≥ 10.
* Peak urinary flow of < 12 ml/sec
* No pathology found with kidney US
* Prostatic urethra length < 30 mm
* Prostate volume < 35 cc
* Normal Urinalysis and urine culture.

Exclusion Criteria:

Main EC:

* Any prior prostate treatment
* Suspected or proved carcinoma of prostate
* Urethral stricture
* Urinary bladder stones
* Serum prostate specific antigen level > 4 ng/ml (unless proved to be carcinoma free by biopsy).
* Active urinary tract infection as determined by positive culture, bacterial prostatitis within the past year documented by positive culture.
* Median prostatic lobe enlargement or a prominent obstructing "ball valve" prostatic lobe.
* Subject has an interest in future fertility and is not willing to undergo fertility treatments whatsoever.
* Any serious medical condition likely to impede successful completion of the study

Intraoperative EC:

* Irregular findings by the implanting physician during the implantation procedure by the cystoscopy that to the best of the implanting physician are exerting non compliance with the exclusion or inclusion criteria and that were not noticed previously during screening

Ages: 50 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Device related and unanticipated SAE | At 3 months
  Device related and unanticipated SAEs will be followed. No such SAEs are expected.

SECONDARY OUTCOMES:
Reduce at least 3 point in the International Prostate Symptom Score (IPSS) in at least 75% of subjects | At 3 months
  Questionnaire of IPSS will be done in each visit.
Increase of maximal urinary peak flow by at least 3 ml/s in at least 75% of subjects | At 3 months
  Maximal uroflow will be measured in each visit

CONTACTS AND LOCATIONS:
Overall Officials: Roy Farfara, MD, Principal Investigator — Bnai Zion Medical Center, Haifa, Israel
Locations (1):
- Meir Medical center, Kfar Saba, Israel